CLINICAL TRIAL: NCT02317770
Title: Comparison of Topical and Nebulized Anesthesia in Patients Undergoing Esophago-Gastro-Duodenoscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SI534/2013
Record Dates: First submitted 2014-12-11; First posted 2014-12-16 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Anesthesia of Mucous Membrane
Keywords: lidocaine, esophago-gastro-duodenoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine Spray (Active Comparator): 20 puffs of 10% Lidocaine spray
  Interventions: Drug: Lidocaine Spray
- Nebulized Lidocaine (Active Comparator): 2.5 mL of 10% Lidocaine
  Interventions: Drug: Nebulized Lidocaine

INTERVENTIONS:
Drug: Lidocaine Spray — 5 puffs of 10% Lidocaine spray is administered every 5 minutes for 4 times. Then the patient is undergone procedure 5 minutes later.
  Other Names: Xylocaine Spray
  Arms: Lidocaine Spray
Drug: Nebulized Lidocaine — The patient receives 2.5 mL of 10% lidocaine is used by nebulizer under oxygen flow 6-7 LPM for 15 minutes prior the procedure.
  Other Names: Nebulized Xylocaine
  Arms: Nebulized Lidocaine

SUMMARY:
This study compares the effect of nebulized lidocaine and lidocaine spray in patients undergoing esophago-gastro-duodenoscopy. The investigators evaluate the success rate of the procedure between two methods.

DETAILED DESCRIPTION:
This is a randomized-controlled trial in the patients undergoing esophago-gastro-duodenoscopy. The patients are randomized by computer into two arms: nebulized lidocaine and lidocaine spray. Both drugs are applied 15-20 minutes prior the prior the procedure. Only one endoscopist participate in this study. After the procedure finishes, the investigators evaluate the outcome and satisfaction of patients and endoscopist.

ELIGIBILITY:
Inclusion Criteria:

* elective case for esophago-gastro-duodenoscopy with ASA classification 1-2
* Both genders
* Age between 18-65 years

Exclusion Criteria:

* History of smoking
* Upper respiratory tract infection
* Asthma
* Heart disease
* Allergy to local anesthetic drugs

Withdrawal or termination criteria

* Patient refusal
* Patient develops lidocaine allergy
* Bronchospasm
* Sign of Local Anesthetic Toxicity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Comparison of Topical and Nebulized Anesthesia | 90 min
  Both nurse anesthetist and endoscopist evaluate difficulty during the procedure and demand for additional sedative drugs using numeric scale

SECONDARY OUTCOMES:
Patient Satisfaction | 90 min
  Satisfaction is evaluated using Numeric Rating Scale (0-10)
Operator Satisfaction | 30 min
  Satisfaction is evaluated using Numeric Rating Scale (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Papiroon Noitasaeng, RN, Principal Investigator — Department of Anesthesia, Faculty of Medicine Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

REFERENCES:
- [Background] Korttila K, Tarkkanen J, Tarkkanen L. Comparison of laryngotracheal and ultrasonic nebulizer administration of lidocaine in local anaesthesia for bronchoscopy. Acta Anaesthesiol Scand. 1981 Apr;25(2):161-5. doi: 10.1111/j.1399-6576.1981.tb01628.x. PMID 7324824
- [Background] Dhir V, Swaroop VS, Vazifdar KF, Wagle SD. Topical pharyngeal anesthesia without intravenous sedation during upper gastrointestinal endoscopy. Indian J Gastroenterol. 1997 Jan;16(1):10-1. PMID 9167371